CLINICAL TRIAL: NCT03157323
Title: Implementing a Low Glycemic Diet in Children and Adolescents Undergoing Treatment for Acute Lymphoblastic Leukemia
Brief Title: Low GI Diet in Children and Adolescents With ALL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Cancer Society, Inc. (Other); Gabrielle's Angel Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ9790
Record Dates: First submitted 2017-04-06; First posted 2017-05-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Obesity, Pediatric
Keywords: Glycemic Index; Acute Lymphoblastic Leukemia; Dietary Change; Pediatric Oncology
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Glycemic Index Diet (Other): Following a low glycemic index diet verses a standard american diet.
  Interventions: Behavioral: Low Glycemic Index Diet

INTERVENTIONS:
Behavioral: Low Glycemic Index Diet — The nutritional intervention is theory-based and will provide nutritional education and counseling to children and their families. Nutritional counseling will be provided by the institutional designate and will focus on increasing patients' understanding of the benefits of a low GI diet, increase knowledge of low GI diet, overcoming barriers, and establishing expectations of the diet.

SUMMARY:
The study aims to determine the feasibility of a 6-month low glycemic dietary intervention in children and adolescents undergoing treatment for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common childhood malignancy with survival exceeding 90%. However, treatment-related toxicity remains a clinical challenge during and after treatment. Evidence-based, nutritional interventions may minimize the development of nutrition-related toxicities, such as bone morbidities, hypertriglyceridemia, and obesity. To date, no effective interventions are available to prevent nutrition-related morbidities in children with ALL. Clinical studies evaluating the glycemic indices in other pediatric conditions have been encouraging. It is plausible that reducing the glycemic indices of diets during cancer treatment may have a profound clinical effect in this vulnerable pediatric population. Prior to the design and implementation of randomized, controlled trials, epidemiological data describing the Glycemic Index (GI) and Glycemic Load (GL) and the association with clinically important outcomes is needed. Additionally, the feasibility of a dietary intervention must also be explored within the setting of pediatric cancer. This study aims to determine the feasibility, measured by compliance to a low-GI diet, of a 6-month low glycemic dietary intervention in children and adolescents undergoing treatment for ALL. The proposed work will be used for the design and implementation of a multi-center nutritional intervention aimed at improving dietary intake during treatment and its effect on clinically important outcomes. Importantly, the information will be used to drive the formation of evidence-based nutritional guidelines for children with cancer, which will expand into the emerging field of individualized medicine for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Lymphoblastic Leukemia (B-Cell, T-Cell, or Mixed Phenotype)
* Within 3 days of starting the induction phase of treatment for Acute Lymphoblastic Leukemia
* Proficient in English or Spanish

Exclusion Criteria:

* Diagnosis of relapsed Acute Lymphoblastic Leukemia
* Not meeting all of the inclusion criteria

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a 6-month low glycemic dietary intervention in children and adolescents undergoing treatment for ALL. | 6 months
  Feasibility will be measured by compliance to a low glycemic index diet, which will be measured via 24 dietary recall, using the Automated Self-Administered 24-Hour Dietary Assessment Tool. A dietary recall will be taken at 7 timepoints from diagnosis to end of treatment; each recall will be defined categorically as high compliance (GI score <55), moderate compliance (GI score 56-69) and low compliance (GI score >70). Change in glycemic index score will show compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ladas, PhD, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walters M, Mowbray C, Jubelirer T, Jacobs S, Kelly KM, Smith K, Yao Y, Jin Z, Ladas EJ. A bilingual dietary intervention early in treatment is feasible and prevents weight gain in childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2021 May;68(5):e28910. doi: 10.1002/pbc.28910. Epub 2021 Feb 15. PMID 33590674